CLINICAL TRIAL: NCT00114101
Title: A Phase III Randomized, Double-Blind Study of Maintenance Therapy With CC-5013 (NSC # 703813) or Placebo Following Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: Lenalidomide in Treating Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00439; NCI-2009-00439 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB 100104/ECOG 100104; CDR0000434845; CALGB-100104 (Other: Alliance for Clinical Trials in Oncology); CALGB-100104 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: DS Stage I Multiple Myeloma; DS Stage II Multiple Myeloma; DS Stage III Multiple Myeloma; Refractory Multiple Myeloma; Smoldering Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Stem Cell Transplantation; Lenalidomide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (melphalan, autologous PBSCT, lenalidomide) (Experimental): Beginning between day 100-110, patients receive lenalidomide PO once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation
- Arm II (melphalan, autologous PBSCT, placebo) (Placebo Comparator): Beginning between day 100-110, patients receive placebo PO once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Placebo Administration

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm I (melphalan, autologous PBSCT, lenalidomide)
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Placebo Administration — Given PO
  Arms: Arm II (melphalan, autologous PBSCT, placebo)

SUMMARY:
This randomized phase III trial studies lenalidomide to see how well it works compared to a placebo in treating patients with multiple myeloma who are undergoing autologous stem cell transplant. Giving chemotherapy before a peripheral blood stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Biological therapies, such as lenalidomide, may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Giving lenalidomide after autologous stem cell transplant may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of CC-5013 (lenalidomide) in prolonging time to disease progression in patients with multiple myeloma after autologous stem cell transplant (ASCT).

SECONDARY OBJECTIVES:

I. To determine if CC-5013 will increase the complete response (CR) rate in patients with multiple myeloma following ASCT.

II. To compare the progression-free survival (PFS) and overall survival (OS) in patients with multiple myeloma who have undergone ASCT and who then are randomized to either CC-5013 or placebo.

III. To determine the feasibility of long-term administration of CC-5013 to multiple myeloma patients who have undergone ASCT.

OUTLINE:

PERIPHERAL BLOOD STEM CELL (PBSC) MOBILIZATION: Mobilization of autologous PBSC will be performed according to institutional guidelines.

AUTOLOGOUS PBSC TRANSPLANTATION (PBSCT): Patients receive melphalan intravenously (IV) over 30-60 minutes on day -2 or -1 or over 2 days on days -3 and -2 or -2 and -1. Patients undergo autologous PBSCT on day 0.

Patients are then randomized to 1 of 2 maintenance treatment arms. (Note: As of 12/17/09, no more patients will be randomized between lenalidomide and placebo. Patients who have not been randomized as of 12/17/09 will be assigned to lenalidomide.)

ARM I: Beginning between day 100-110, patients receive lenalidomide orally (PO) once daily.

ARM II: Beginning between day 100-110, patients receive placebo (PO) once daily.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have active multiple myeloma requiring treatment (Durie-Salmon stage >= 1) and have stable disease or be responsive to at least 2 months of any induction therapy; patients with smoldering myeloma are not eligible unless the disease has progressed to >= stage 1
* No more than 12 months of any prior therapy, including CC-5013 and thalidomide
* Within 12 months of initiation of induction therapy
* No prior progression after initial therapy; in addition, no more than two regimens will be allowed excluding dexamethasone alone
* No prior peripheral blood, bone marrow, or solid organ transplant
* Patients must have peripheral blood stem cell collection of >= 2 x 10^6 cluster of differentiation (CD)34+ cells/kg (patient body weight) and preferably 5 x 10^6 cells/kg (patient body weight); stem cells may be collected at any time prior to transplant; peripheral blood stem cell collection may occur before or after registration
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have diffusing capacity of the lung for carbon monoxide (DLCO) > 50% predicted with no symptomatic pulmonary disease
* Patients must have left ventricular ejection fraction (LVEF) >= 40% by multi gated acquisition scan (MUGA) or echocardiogram
* Patients must not have uncontrolled diabetes mellitus
* Patients must not have an active serious infection
* Patients must not be human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSag), or hepatitis (Hep) C positive
* Patients must be non-pregnant and non-nursing; women of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL 10-14 days prior to registration and repeated within 24 hours prior to the first dose of lenalidomide; in addition, women of childbearing potential taking lenalidomide must have a pregnancy test performed by the doctor weekly during the first 4 weeks of treatment, and then every 4 weeks if menses are regular and every 2 weeks if menses are irregular, and then 30 days following the last dose of lenalidomide; women of childbearing potential must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control - one highly effective method (intrauterine device [IUD], hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (latex condom, diaphragm, or cervical cap) - at the same time, at least 4 weeks before she begins lenalidomide therapy; "women of childbearing" potential is defined as a sexually mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months; men must agree not to father a child and must use a latex condom during any sexual contact with women of childbearing potential while taking lenalidomide and for 4 weeks after therapy is stopped, even if they have undergone a successful vasectomy
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 100,000/uL
* Creatinine clearance* >= 40 cc/min

  * To be calculated by method of Cockcroft-Gault or after 24-hour urine collection
* Creatinine =< 2 mg/dL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) =< 3 x upper limits of normal
* Alkaline phosphatase =< 3 x upper limits of normal
* Urine (U)-human chorionic gonadotropin (HCG) or serum HCG negative (if patient of childbearing potential)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2004-12-15 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L McCarthy, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (140):
- United States (140):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Centerpoint Medical Center LLC, Independence, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health NCORP, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin

REFERENCES:
- [Derived] Holstein SA, Jung SH, Richardson PG, Hofmeister CC, Hurd DD, Hassoun H, Giralt S, Stadtmauer EA, Weisdorf DJ, Vij R, Moreb JS, Callander NS, van Besien K, Gentile TG, Isola L, Maziarz RT, Bashey A, Landau H, Martin T, Qazilbash MH, Rodriguez C, McClune B, Schlossman RL, Smith SE, Hars V, Owzar K, Jiang C, Boyd M, Schultz C, Wilson M, Hari P, Pasquini MC, Horowitz MM, Shea TC, Devine SM, Linker C, Anderson KC, McCarthy PL. Updated analysis of CALGB (Alliance) 100104 assessing lenalidomide versus placebo maintenance after single autologous stem-cell transplantation for multiple myeloma: a randomised, double-blind, phase 3 trial. Lancet Haematol. 2017 Sep;4(9):e431-e442. doi: 10.1016/S2352-3026(17)30140-0. Epub 2017 Aug 17. PMID 28826616
- [Derived] McCarthy PL, Owzar K, Hofmeister CC, Hurd DD, Hassoun H, Richardson PG, Giralt S, Stadtmauer EA, Weisdorf DJ, Vij R, Moreb JS, Callander NS, Van Besien K, Gentile T, Isola L, Maziarz RT, Gabriel DA, Bashey A, Landau H, Martin T, Qazilbash MH, Levitan D, McClune B, Schlossman R, Hars V, Postiglione J, Jiang C, Bennett E, Barry S, Bressler L, Kelly M, Seiler M, Rosenbaum C, Hari P, Pasquini MC, Horowitz MM, Shea TC, Devine SM, Anderson KC, Linker C. Lenalidomide after stem-cell transplantation for multiple myeloma. N Engl J Med. 2012 May 10;366(19):1770-81. doi: 10.1056/NEJMoa1114083. PMID 22571201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2004 and July 2009, a total of 568 participants were recruited to this study.
Pre-assignment Details: After registration, participants underwent a peripheral blood stem cell transplant. Of the 568 participants, 460 were randomized to either arm, stratified by beta2 microglobulin, prior thalidomide use and prior lenalidomide use. (108 participants dropped out prior to randomization, most common reasons include: progression, ineligible, refusal)
Groups:
- Lenalidomide Maintenance: Beginning between day 100-110, patients receive oral lenalidomide once daily - 10 mg/day for the first 3 months, then if tolerated, 15 mg/day.
- Placebo Maintenance: Beginning between day 100-110, patients receive oral placebo once daily - 10 mg/day for the first 3 months, then if tolerated, 15 mg/day.
  (closed as of 12/17/09)
Period: Overall Study
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Started | 231 | 229
Completed | 231 | 229
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance | Total
Number analyzed (Participants) | 231 | 229 | 460
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 71] | 58 [40 to 71] | 59 [29 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 100 | 210
  Male | 121 | 129 | 250
Region of Enrollment [Number; unit: participants]
  United States | 231 | 229 | 460
Beta 2 microglobulin at registration [Number; unit: participants]
  > 2.5 mg/liter | 50 | 55 | 105
  <= 2.5 mg/liter | 170 | 163 | 333
  Missing data | 11 | 11 | 22
Prior use of thalidomide during induction [Number; unit: participants]
  Yes | 102 | 103 | 205
  No | 129 | 126 | 255
Prior use of lenalidomide during induction therapy [Number; unit: participants]
  Yes | 79 | 81 | 160
  No | 152 | 148 | 300

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the date of transplant to date of progression or death due to any cause, whichever occurs first. TTP was estimated using the Kaplan Meier method.
  Progression was defined per the International Myeloma Working Group definition as one more of the following:
  * 25% increase in serum M-component (absolute increase >= 0.5g/dl)
  * 25% increase in urine M-component (absolute increase >= 200mg/24hour
  * 25% increase in the difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl)
  * 25 % increase in bone marrow plasma cell percentage (absolute increase of >=10%)
  * Definite development of new bone lesion or soft tissue plasmacytomas
  * Development of hypercalcemia
Time Frame: Duration of study (up to 10years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Number analyzed (Participants) | 231 | 229
months | 39 [36 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 21 [18 to 28]
Statistical Analysis 1: Comparison: Lenalidomide Maintenance vs Placebo Maintenance; Test type: Non-Inferiority or Equivalence — This study was designed to have 80% power, with the use of the log-rank test at a one-sided significance level of 0.05, to detect a hazard ratio of 1.4, assuming proportional hazards and an exponential time to event distribution. Under the assumed framework, 309 events were expected. The expected drop out rate before randomization was 15%; p < 0.001, Log Rank — Participants were randomized with the use of a permuted-block design stratified by beta 2 microglobulin, prior use of thalidomide and prior use of lenalidomide. TTP was monitored with the use of a group sequential design for superiority and futility; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.26 to 0.53]

2. Secondary Outcome: Response to Autologous Hematopoietic Stem-cell Transplant (HSCT) at Day 100
Description: Response was defined according to International Myeloma Working Group criteria (2006)
  * Complete Response: Complete disappearance of M-protein from serum & urine on immunofixation, normalization of Free Light Chain (FLC) ratio & <5% plasma cells in bone marrow (BM)
  * Partial Response: >= 50% reduction in serum M-Component and/or Urine M-Component >= 90% reduction or <200 mg per 24 hours; or >= 50% decrease in difference between involved and uninvolved FLC levels
  * Marginal Response: 25-49% reduction in serum M-component & urine M-component by 50-89% which still exceeds 200mg/24hour
  * Progressive Disease: Defined in primary outcome measure
  * Stable Disease: Not meeting any of the criteria above
Time Frame: Day 100
Measure: Number; unit: participants
Groups:
- Lenalidomide Maintenance: Beginning between day 100-110, patients receive oral lenalidomide once daily.
- Placebo Maintenance: Beginning between day 100-110, patients receive oral placebo once daily.
  (closed as of 12/17/09)
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Number analyzed (Participants) | 231 | 229
participants
  Complete response | 67 | 79
  Partial response | 115 | 109
  Marginal response | 11 | 5
  Stable disease | 38 | 32
  Progressive disease | 0 | 3
  Unknown | 0 | 1

3. Other Pre Specified Outcome: Overall Survival
Description: Overall Survival was measured from the date of randomization to date of death due to any cause. OS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Number analyzed (Participants) | 231 | 229
months | NA [NA to NA] — The median overall survival has not been reached. | NA [NA to NA] — The median overall survival has not been reached.
Statistical Analysis 1: Comparison: Lenalidomide Maintenance vs Placebo Maintenance; Test type: Superiority or Other; p = 0.70, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.26 to 1.02]

4. Post Hoc Outcome: Number of Participants With Progression, Death or Diagnosis of Second Primary Malignancy
Description: Patients who develop progression (defined in primary outcome measure), died or develop a new primary malignancy (cancer) will summarized in this outcome.
Time Frame: Duration of study (up to 10 years)
Measure: Number; unit: participants
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Number analyzed (Participants) | 231 | 229
participants | 92 | 133
Statistical Analysis 1: Comparison: Lenalidomide Maintenance vs Placebo Maintenance; Test type: Superiority or Other; p < 0.001, Fisher Exact; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.41 to 0.69]

ADVERSE EVENTS:
Arm/Group | Lenalidomide Maintenance | Placebo Maintenance
Serious Adverse Events (participants affected / at risk) | 52/231 | 33/229
Other Adverse Events (participants affected / at risk) | 195/231 | 166/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide Maintenance (N=231) | Placebo Maintenance (N=229)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 8 (8) | 5 (5)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Thyroid function high (hyperthyroidism thyrotoxicosis) (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 19 (22) | 9 (9)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Obstruction GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ulcer, GI (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constitutional Symptoms - Other (General disorders) | 0 (0) | 2 (2)
Death not associated with CTCAE term (General disorders) | 2 (2) | 2 (2)
Edema: limb (General disorders) | 1 (1) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3) | 2 (2)
Fever (General disorders) | 3 (3) | 4 (4)
Pain - Other (General disorders) | 1 (1) | 2 (2)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 16 (18) | 7 (7)
Infection - Other (Infections and infestations) | 4 (4) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 14 (14) | 9 (13)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 7 (8)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 (3) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 (4) | 1 (1)
Alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 10 (12) | 4 (5)
Cardiac troponin I (cTnI) (Investigations) | 0 (0) | 1 (1)
Creatinine (Investigations) | 1 (2) | 3 (3)
Fibrinogen (Investigations) | 0 (0) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 2 (2) | 1 (1)
Leukocytes (total WBC) (Investigations) | 10 (11) | 2 (2)
Lipase (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 5 (5) | 3 (3)
Metabolic/Laboratory - Other (Investigations) | 1 (1) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 40 (47) | 14 (16)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 1 (1)
Platelets (Investigations) | 39 (45) | 16 (21)
Weight gain (Investigations) | 1 (1) | 3 (3)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Magnesium serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 9 (12)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mental status (Nervous system disorders) | 1 (1) | 0 (0)
Neurology - Other (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Mood alteration (Psychiatric disorders) | 4 (4) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2) | 2 (3)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (5)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide Maintenance (N=231) | Placebo Maintenance (N=229)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (10) | 3 (4)
Hemoglobin (Blood and lymphatic system disorders) | 26 (45) | 9 (22)
Hemolysis (e.g. immune hemolytic anemia drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 1 (1)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 1 (1) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid function high (hyperthyroidism thyrotoxicosis) (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (2) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 0 (0) | 4 (4)
Vision-blurred vision (Eye disorders) | 1 (1) | 1 (2)
Watery eye (epiphora tearing) (Eye disorders) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (10) | 7 (12)
Dental: periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 89 (227) | 52 (90)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (2) | 3 (4)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 3 (3) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melena/GI bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (15) | 10 (15)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies if specified in the protocol. (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (10) | 6 (9)
Constitutional Symptoms - Other (General disorders) | 0 (0) | 2 (2)
Edema: limb (General disorders) | 4 (5) | 3 (3)
Edema:head and neck (General disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 36 (55) | 29 (54)
Fever (General disorders) | 9 (10) | 2 (2)
Flu-like syndrome (General disorders) | 1 (1) | 0 (0)
Pain - Other (General disorders) | 1 (1) | 8 (14)
Rigors/chills (General disorders) | 4 (6) | 1 (3)
Syndromes - Other (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Allergy/Immunology - Other (Immune system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 16 (17) | 11 (14)
Infection - Other (Infections and infestations) | 6 (6) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 11 (14) | 14 (18)
Infection with unknown ANC (Infections and infestations) | 15 (18) | 9 (11)
Infection without neutropenia (Infections and infestations) | 2 (3) | 1 (1)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (1) | 1 (1)
Viral hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intra-operative injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 11 (13) | 2 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 7 (8) | 3 (5)
Alkaline phosphatase (Investigations) | 5 (5) | 4 (4)
Bilirubin (hyperbilirubinemia) (Investigations) | 24 (66) | 18 (36)
CPK (creatine phosphokinase) (Investigations) | 1 (3) | 0 (0)
Creatinine (Investigations) | 2 (2) | 5 (9)
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 0 (0) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 3 (7) | 0 (0)
Leukocytes (total WBC) (Investigations) | 29 (72) | 14 (33)
Lymphopenia (Investigations) | 17 (31) | 9 (23)
Metabolic/Laboratory - Other (Investigations) | 2 (3) | 3 (4)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 153 (593) | 75 (181)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 2 (2)
Platelets (Investigations) | 129 (445) | 78 (200)
Weight gain (Investigations) | 13 (21) | 21 (33)
Weight loss (Investigations) | 1 (2) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 6 (7)
Calcium serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Calcium serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 (6) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 (12) | 7 (18)
Glucose serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Phosphate serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Potassium serum-low (hypokalemia) (Metabolism and nutrition disorders) | 9 (11) | 4 (7)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Triglyceride serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Uric acid serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 35 (84) | 50 (154)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (8) | 8 (9)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage CNS (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1) | 4 (4)
Neuropathy: cranial (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 6 (10) | 4 (6)
Neuropathy: sensory (Nervous system disorders) | 24 (40) | 24 (49)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (dysgeusia) (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (15)
Libido (Psychiatric disorders) | 1 (1) | 1 (1)
Mood alteration (Psychiatric disorders) | 9 (12) | 11 (16)
Hemorrhage GU (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 3 (3) | 3 (3)
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 (1) | 3 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3) | 4 (4)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergic rhinitis (including sneezing nasal stuffiness postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (7)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 9 (13)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (8)
Hemorrhage pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (12)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 57 (86) | 36 (56)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (5)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (hives welts wheals) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Hemorrhage/Bleeding - Other (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less